CLINICAL TRIAL: NCT00970528
Title: A Randomized, Parallel Group, Open-Label, Active-Controlled Study Comparing Acarbose With Voglibose in Patients Who Are Inadequately Controlled With Insulin Glargine Alone or in Combination With Metformin Based on Glycemic Control
Brief Title: Glucose Reduction by Early Acarbose Treatment in Basal Insulin
Acronym: GREAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14081
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Oral Hypoglycemic Agent
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acarbose; voglibose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Acarbose (Glucobay, BAYG5421)
- Arm 2 (Active Comparator)
  Interventions: Drug: Voglibose (Basen)

INTERVENTIONS:
Drug: Acarbose (Glucobay, BAYG5421) — uptitrated 100mg three times a day with insulin glargine alone or in combination with metformin
  Arms: Arm 1
Drug: Voglibose (Basen) — uptitrated 0.3mg three times a day with insulin glargine alone or in combination with metformin
  Arms: Arm 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of acarbose in comparison with voglibose in type 2 diabetic patients whose blood glucose levels were inadequately controlled with insulin glargine alone or in combination with metformin.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-79 years
* Type 2 diabetes inadequately controlled with insulin glargine alone or in combination with metformin

  * Diagnosed of type 2 diabetes for at least 6 months prior to screening
  * Treated with tolerable, stable dose of insulin glargine and/or metformin for at least 3 months prior to screening
  * HbA1C > 7.0 and </= 10.0% at screening

Exclusion Criteria:

* Type 1 diabetes patients
* Myocardial infarction, unstable angina or coronary artery bypass surgery within previous 6 months
* Clinical evidence of active liver disease, or serum ALT or AST 3 times the upper limit of the normal (ULN) range
* Serum creatinine >/= 1.5 mg/dl for males, >/= 1.4 mg/dl for females
* Active proliferative diabetic retinopathy
* Any other anti-diabetic medications except insulin glargine and metformin within 4 weeks prior to study entry
* Gastrointestinal diseases that are likely to be associated with abnormal intestinal motility or altered absorption of nutrients (e.g. gastroparesis, malabsorption syndrome, chronic diarrhea states, enteropathies, inflammatory bowel disease, partial intestinal obstruction, and large hernias)
* Galactose intolerance
* Pregnancy
* Delivery, abortion, or lactation within less than three cycles before the start of treatment
* No use of contraceptive in childbearing aged. Women of childbearing potential must agree to use adequate contraception (barrier method of birth control) since signing of the informed consent form until at least 30 days after the last study drug administration.
* Hypersensitivity to the active substances or any of gradient of the study drug ingredients
* Treatment with any medication including corticosteroid or herb medication that can affect blood glucose level in the 3 months prior to study entry
* Any disease or condition that in the opinion of the investigator may interfere with completion of the study

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2009-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Glycosylated hemoglobin (HbA1c) | Change from baseline to week 24, at week -2, 0, 8 and 24

SECONDARY OUTCOMES:
Self monitoring blood glucose concentration | 6 points for 2 days prior to each visit (at week 0, 4, 8, 16 and 24)
Fasting blood glucose concentration | At week -2, 0, 4, 8, 16 and 24
Blood concentration of triglyceride | At week -2 and 24
Blood concentration of low density lipoprotein | At week -2 and 24
Blood concentration of total cholesterol | At week -2 and 24
Blood concentration of high density lipoprotein | At week -2 and 24
Blood concentration of apolipoprotein A-1 | At week -2 and 24
Blood concentration of apolipoprotein B | At week -2 and 24
Blood concentration of Glucagon-like peptide-1 (GLP-1) | At week -0 and 24
Body weight, Body Mass Index(BMI) | At week -2, 0, 4, 8, 16 and 24
High Sensitivity C-reactive protein (hs-CRP) | At week -2 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (9):
- South Korea (9):
  - Wŏnju, Gang''weondo
  - Busan, Korea
  - Gyeonggi-do, Korea
  - Pusan, Korea
  - Seoul, Korea
  - Daegu
  - Jeonju
  - Seongbuk-gu Seoul
  - Seoul

REFERENCES:
- [Derived] Lee MY, Choi DS, Lee MK, Lee HW, Park TS, Kim DM, Chung CH, Kim DK, Kim IJ, Jang HC, Park YS, Kwon HS, Lee SH, Shin HK. Comparison of acarbose and voglibose in diabetes patients who are inadequately controlled with basal insulin treatment: randomized, parallel, open-label, active-controlled study. J Korean Med Sci. 2014 Jan;29(1):90-7. doi: 10.3346/jkms.2014.29.1.90. Epub 2013 Dec 26. PMID 24431911